CLINICAL TRIAL: NCT04574778
Title: Randomized Trial of IV Versus Oral Acetaminophen for Ambulatory Lumbar Discectomy or Single-level Decompression
Brief Title: Randomized Trial of Intraoperative IV Versus Preoperative Oral Acetaminophen During Ambulatory Lumbar Discectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GSCHR19D.660
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative; Spine Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only those performing postoperative assessments and the participants will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: IV acetaminophen and PO placebo (Active Comparator): Group 1 will receive 1000 mg of IV acetaminophen approximately 30 minutes prior to skin closure and will receive oral placebo in the holding area prior to surgery
  Interventions: Drug: Acetaminophen
- Group 2: PO acetaminophen (Active Comparator): Group 2 will receive 1000 mg of PO acetaminophen in the holding area and will not receive an IV placebo.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — 1000 mg of oral acetaminophen preoperatively administered

SUMMARY:
Effective non-opioid analgesics are of particular interest in ambulatory surgery, as providers may be able to reduce pain while avoiding perioperative opioids that can delay same day discharge. The value of maintaining an efficient flow of patients from the perioperative area to discharge is an important metric for same day surgery centers, and an improvement in efficiency with IV acetaminophen could potentially offset the increased cost of the medication while providing a more pleasant surgical experience for patients. The goal of this study is to compare the efficacy of intraoperative IV administration vs. preoperative oral administration of acetaminophen on postoperative opioid utilization, patient-reported pain scores, opioid-related adverse effects, and time to recovery and discharge from the post-anesthesia care unit (PACU) after ambulatory lumbar discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years-old
* Weight greater than 50 kg body weight
* ASA physical status I-III
* English-speaking

Exclusion Criteria:

* Weight less than 50 kg
* Pregnancy or breast feeding
* revision surgery
* Contraindications to the administration of acetaminophen (e.g. allergy, liver failure, etc)
* Chronic pain conditions unrelated to back pain
* Opioid tolerance ( defined as taking greater than oxycodone 20 mg daily for a week during the past month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid usage | 1 day
  Postoperative opioid usage over the first 24 hours will be reported in IV morphine equivalents

SECONDARY OUTCOMES:
Quality of recovery | 1 day
  assessed using the Quality of Recovery 15 scale, with a range of 0-150 (0 is the worst score and 150 is the best possible recovery)
Number of patients who report nausea or vomiting | 1 day
  this will be a count of the number of patients who report nausea or vomiting in recovery room
Mean pain score | 1 day
  (0-10 numerical rating scale where 0=no pain and 10=worst pain imaginable) - this will be the mean pain rating upon entering pacu and at least 1 other time point in each study group

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwenk ES, Ferd P, Torjman MC, Li CJ, Charlton AR, Yan VZ, McCurdy MA, Kepler CK, Schroeder GD, Fleischman AN, Issa T. Intravenous versus oral acetaminophen for pain and quality of recovery after ambulatory spine surgery: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jun 10;50(6):483-488. doi: 10.1136/rapm-2024-105386. PMID 38499358